CLINICAL TRIAL: NCT01846780
Title: The Effect of PTA & Stenting on Intravenous Pressure in Deep Venous Obstructive Disease Before, After and During Ambulation on a Treadmill - Pilot Study.
Brief Title: Treadmill Pilot Study (Invasive Pressure Measurements in PTS)
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL44588
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Post-thrombotic Syndrome; May-Thurner Syndrome
MeSH Terms: conditions — Postthrombotic Syndrome; May-Thurner Syndrome | interventions — Stents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for possible future research
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Venous outflow obstruction lower limb: Patients with unilateral post-thrombotic iliac vein/common femoral vein obstruction undergoing PTA & stenting (possibly with additional endophlebectomy and AV-fistula)
  Interventions: Procedure: PTA & stenting

INTERVENTIONS:
Procedure: PTA & stenting — PTA & stenting of the iliac veins and/or common femoral vein. Patients who need to undergo endophlebectomy of the common femoral vein with AV-fistula creation are also included.

SUMMARY:
Patients with unilateral post-thrombotic obstruction of the iliac tract and or common femoral vein, eligible for stenting are included. Intravenous pressure is measured in both dorsal foot veins and both common femoral veins. Patients are asked to undergo a standardised treadmill test (3.2km/h, 0% slope that increases by 2%/2min, maximum walking time 26 min). Painfree and maximum action radius are noted.

DETAILED DESCRIPTION:
Rationale: PTA & stenting in iliofemoral and iliocaval venous obstruction has been proven to be an effective method of treatment with good clinical results. However, no proper investigations have been made to objectify the reduction in (ambulatory) venous hypertension caused by this type of obstruction. Normal ambulatory venous pressure is below 20mmHg, though studies have already shown a linear relationship between the incidence of ulcers and an ambulatory intravenous pressure of more than 30mmHg. We believe that by measuring the (ambulatory) venous pressure before and after stenting, we will gain more knowledge on the hemodynamics of venous disease and its treatment and we will obtain information that might identify patients at risk of stent occlusion or the forming of an ulcer in an early stage. Identifying these patients will most certainly influence preventive treatment in the future.

Objective: To map the changes in intravenous pressure in post-thrombotic iliofemoral venous obstruction and evaluate the effect of PTA & stenting with possible identification of a predictive parameter for success of treatment.

Study design: Prospective, observational study (healthy and diseased limb in one patient).

Study population: Patients with an iliofemoral venous obstruction, objectified on duplex ultrasonography and magnetic resonance venography, and the indication for stenting of the obstructed tract(s).

Intervention: All patients will undergo stenting of the obstructed venous tract. Patients receive the same therapy as they would have received not participating in this study; therefore this study has no influence on the treatment patients receive.

Main study parameters/endpoints: Primary outcome is the change in (ambulatory) venous pressure after stenting for deep venous obstructive disease. Other important endpoints are the absolute values for intravenous pressure, pain free walking distance and maximum walking distance. Additional outcome measurements are stent patency, CEAP score, Villalta score, venous clinical severity score, and generic and disease specific quality of life scores. Finally, transverse surface area, diameter and circumference of the common femoral vein will be measured.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients have to make three visits. Each visit will take approximately two hours. During each test day, patients will undergo intravenous pressure measurements in both dorsal foot veins, both common femoral veins and a vein in the left upper arm, which are measured via a venflon needle or microsheath (placed under ultrasound guidance) connected to a pressure transducer; a treadmill test lasting maximally 26 minutes; an air plethysmography, which they need to undergo anyway; and a duplex ultrasound to assess the common femoral vein. This is a very low risk study, since all diagnostic tools that are used or also used in usual clinical practice and given the low risk on mild complications. Patients can experience pain due to the insertion and removal of the venflons/microsheaths, due to compression of the groin after removal of the microsheaths and due to walking on a treadmill (because of venous claudication).

Amendment:

iv in the arm vein as a control is not performed anymore. An abdominbal wall collateral is cannulated instead, if present.

ELIGIBILITY:
Inclusion Criteria:

* Indication for stenting (possibly with endophlebectomy and AV-fistula), minimally 18 years of age, life expectancy of at least 6 months.

Exclusion Criteria:

* Younger than 18 years of age, life expectancy of less than 6 months, venous obstruction in the contralateral limb, peripheral arterial disease, pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at our specialized venous outpatient clinic in our tertiary centre
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change in (ambulatory) venous pressure | 0 months, 3months
  measured at the dorsal foot vein and common femoral vein

SECONDARY OUTCOMES:
VCSS | 0 months, 3months
Villalta scale | 0 months, 3months
Quality of Life | 0 months, 3months
Patency | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cees Wittens, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Kurstjens RL, de Wolf MA, Konijn HW, Toonder IM, Nelemans PJ, de Graaf R, Wittens CH. Intravenous pressure changes in patients with postthrombotic deep venous obstruction: results using a treadmill stress test. J Thromb Haemost. 2016 Jun;14(6):1163-70. doi: 10.1111/jth.13333. Epub 2016 May 31. PMID 27061685